



# Statistical Analysis Plan Checklist for Investigator Initiated Trials

Open-Label Study to Determine the Feasibility of MLN9708 as Maintenance after Allogeneic Stem Cell Transplant for Multiple Myeloma, Followed by an Expansion Phase at the Maximum-Tolerated Dose (MTD)

Sponsor: Sarah Cannon Development Innovations

(Innovations)

Study Drug: MLN9708

SCRI Protocol Number: MM 42

REFERENCE SOP: CDS-0102

Prepared By: Innovations

Version 1.0, 06 JAN 2020 






REFERENCE SOP: CDS-0102 Template ID: ASSOC-DOC-116-SOP [B] Confidential




REFERENCE SOP: CDS-0102

# Statistical Analysis Plan Checklist for Investigator Initiated Trials History of Changes

This document has undergone the following changes:

| Version Number | Version Date | Description of Changes |
|----------------|--------------|------------------------|
| 1.0 | 06 JAN 2020 | Original document |







REFERENCE SOP: CDS-0102

### Statistical Analysis Plan Checklist Review and Approval

| Approved By: | |
|----------------------------------------------|------|
| Innovations<br>Biostatistician<br>David Bass | Date |
| Innovations<br>Managerial Peer-Reviewer | Date |
| Innovations Tion 1 Manager | Date |
| Innovations Study Chair | Date |






| 1.1 Objectives | |
|---|---|
| Primary Objective: | Safety of MLN9708 when used as maintenance after allogeneic stem cell transplant for multiple myeloma |
| Secondary Objectives: | Maximum-tolerated dose (MTD) of MLN9708 in this patient population |
| | Progression-free survival (PFS) at 2 years after initiation of maintenance therapy |
| | Overall survival (OS) at 2 years after allogeneic stem cell transplant |
| | Incidence of graft-versus-host disease (GVHD) in patients receiving allogeneic stem cell transplant and maintenance with MLN9708 |
| | Effect of MLN9708 on immune effector cells after allogeneic stem cell transplant |
| 1.2 Study Design | |
| Study Type | ⊠ Non-Randomized |
| | ☐ Randomized (Allocation Ratio: ) |
| Details | This is a Phase II, open-label, multicenter, non-randomized study to determine the feasibility of MLN9708 as maintenance after allogeneic stem cell transplant for multiple myeloma. Patients will be enrolled between Days 45 and 120 after allogeneic transplant and will receive MLN9708 on Days 1, 8, and 15 of each 28-day cycle for 6 cycles. Up to 18 patients will be enrolled in the dose-escalation phase to define the MTD of MLN9708. An additional 20 patients will be enrolled in the expansion phase at the MTD. |
| | PFS is defined as the time from the first day of study drug administration (Day 1) to disease progression as defined by the International Myeloma Working Group Uniform Response Criteria (see Appendix E of protocol), or death on study. Patients who are alive and free from disease progression will be censored at the date of last tumor assessment. |
| | OS is defined as the time from the first day of study drug administration (Day 1) to death on study. Patients who are alive will be censored at the date of last known date alive. |
| | PFS and OS (efficacy secondary endpoints) estimates will be generated using Kaplan-Meier methods, both for all patients enrolled and those patients receiving the MTD. Two-year PFS and OS estimates with 95% confidence intervals (CIs), and median PFS and OS with 95% CIs, will be generated and reported accordingly. |
| 1.3.2 Randomization | |
| Randomization Type: | ☐ Open-Label ☐ Single Blind ☐ Double-Blind |
| 1.4 Timing of Analysis | |
| Planned Interim Analysis | ⊠ Cohort Review / Dose Escalation |
| | ⊠ Safety Review |
| | ☐ Interim Efficacy/Safety Analysis |
| | ☐ Independent DMC/DSMB |
| | ☐ Annual Report / Investigator Brochure (IB) |
| | ☐ Abstract / Scientific Presentation (Oral/Poster) |
| Final Analysis | As determined by the Study Chair in consultation with the clinical team |






REFERENCE SOP: CDS-0102

| 1.5 Responsibilities | |
|---|---|
| Trial Statistician: | Prepare SAP checklist and TFL shells. Review deliverables produced by Statistical Programmers. |
| PK Statistician: | N/A |
| Independent Statistician: | N/A |
| 1.6 Analysis Software | |
| Main statistical analysis: | SAS Version 9.3 or above |
| Other analysis software: | N/A |






| 1.7 Coding | |
|---|---|
| <ul><li>☑ Adverse Events</li><li>☐ Medical History</li></ul> | <ul> <li>✓ MedDRA:</li></ul> |
| ☐ Concomitant Medication ☐ Prior Therapy ☐ Subsequent/Further Therapy | ☐ WHO-Drug: ☐ Version ☐ Most current release and update coding with new major releases |
| 3 Analysis Population | |
| Intent-To-Treat (ITT) Population definition: | <ul> <li>☐ All patients who have started treatment in the study</li> <li>☐ All patients who have been randomized in the study, regardless of whether they have received any treatment or not</li> <li>☐ All patients who have been randomized and have started treatment in the study</li> <li>☐ Other definition, specify:</li> </ul> |
| Per Protocol (PP) Population to be used in analysis: | ☐ Yes ☐ No If yes, please specify the criteria for exclusion from the PP population: |
| Safety (SAF) Population definition | <ul><li>☑ The Safety population will consist of all patients who received at least one dose of MLN9708.</li><li>☐ Other definition, specify:</li></ul> |
| Other Analysis Population definition: | The Efficacy Evaluable population will consist of all patients with measurable or evaluable disease at baseline who receive at least 1 dose of MLN9708 and undergo at least one post-baseline disease assessment. In addition, patients who discontinued the study prior to their first post-baseline disease assessment due to death or progressive disease will also be included in the Efficacy Evaluable population. |
| 4 Baseline Value Definitions | |
| | Information collected and procedures performed for each patient at ≤7 days prior to initiation of treatment. |
| 5/6 Efficacy | |
| Response Criteria Used: | <ul> <li>□ RECIST 1.0</li> <li>□ RECIST 1.1</li> <li>□ Cheson 2007</li> <li>□ Modified RECIST – specify:</li> <li>□ Other criteria, Specify:</li> <li>International Myeloma Working Group Uniform Response Criteria</li> </ul> |
| Efficacy Assessment Timepoints: | Patients will be re-evaluated for response to treatment after 2 cycles of treatment. Response will be assessed at 8-week intervals (±1 week) during study treatment. Patients with progressive disease (PD) or unacceptable toxicity should be discontinued from the study; patients with stable disease (SD) or response to therapy will continue treatment through 6 cycles. |






| Efficacy Endpoints: | | | 1 | | |
|---|---|---|---|---|---|
| | | Endpoint | Primary Analysis<br>Population | Other Anal<br>Population | |
| | Primary | PFS | Efficacy Evaluable | | |
| | Secondary | os | Efficacy Evaluable | | |
| Definition of Terms: | | | | | |
| ⊠ Response | | Response + Partial Resp | | - | |
| | | Response + Partial Resp | onse, confirmed with | weeks | apart. |
| | ⊠ Other crit<br>Internat | ena, specify:<br>ional Myeloma Working G | roup Uniform Response | e Criteria: | |
| | VGPR (ver | VGPR (very good partial response) PR (partial response) | | | |
| ☐ Clinical Benefit | ☐ Complete Response + Partial Response + Stable Disease as best observed response | | | | |
| | Complete Response + Partial Response (confirmed with Stable Disease (at least weeks from start of treatment) weeks apart) + | | | | |
| | Other criteria, specify: | | | | |
| ⊠ Progression | As reported by Investigator | | | | |
| ☐ Subsequent Therapy | | | | | |
| ☐ Treatment Failure | | | | | |
| Definition of Endpoints: | Start Date: [ | ☐ Date of Randomization | ☑ Date of First T | reatment | |
| | End Date (sp | pecify for all pertinent endp | ooints): | | |
| | Progression-Free Survival: Event = Progression or Death | | | | |
| | | Situation | Date of Event or | | Outcome |
| | No baseline | | Date of first treat | | Censored |
| | | ited between scheduled visit<br>and received no subsequent | ss, First date of evaluation overall response | | Event |
| | did not die, | ited between scheduled visit<br>out received subsequent the<br>rring progression event | | to start of | Censored |
| | | on-study without previous P<br>I no subsequent therapy | Date of death | | Event |
| | | on-study and had previous F<br>I no subsequent therapy | PD, First date of evaluation overall response | | Event |




#### MM 42 Statistical Analysis Plan Checklist

| | Death while on-study without previous PD, but received subsequent therapy prior to death event | Date of last evaluable tumor assessment prior to start of subsequent therapy | Censored |
|---|---|---|---|
| | Death while on-study and had previous PD,<br>but received subsequent therapy prior to PD<br>event | Date of last evaluable tumor assessment prior to start of subsequent therapy | Censored |
| | No progression, no death | Date of last evaluable tumor assessment | Censored |
| | Treatment discontinuation for adverse event or other non-event reason | Date of last evaluable tumor assessment | Censored |
| | Overall Survival: Event = Death | | |
| | Situation | Date of Event or Censoring | Outcome |
| | Death, while on-study or follow-up | Date of death | Event |
| | Alive, as of end of study or follow-up | Date last known alive | Censored |
| | Status unknown, as of end of study | Date last known alive | Censored |
| ☐ Overall Response Rate (ORR) | Default: Estimates of rates in each treatment | t arm | |
| ☐ Disease Control Rate (DCR) | ☐ Difference in rates & 95% confidence inte | erval between treatment arms | |
| ☐ Clinical Benefit Rate (CBR) | D p-value, specify statistical test. | | |
| ☐ Early Progression Rate (EPR) | | | |
| ☐ Time To Progression (TTP) | Default: Estimates of medians in each treatment arm | | |
| □ Progression-Free Survival (PFS) | | | |
| ☑ Overall Survival (OS) | Hazard ratio & 95% confidence interval between treatment arms, unstratified | | |
| , , | ☐ p-value, specify statistical test: ☐ Hazard ratio & 95% confidence interval between treatment arms, stratified (specify | | |
| ☐ Duration of Response | stratification factor(s)): | | |
| ☐ Duration of Stable Disease | p-value, specify statistical test: | | |
| ☐ Time To Treatment Failure (TTF) | | | |
| ☐ Other, Specify: | | | |
| 7 Safety | | | |
| Adverse Events | Definition of Treatment-Emergent Adverse E<br>Treatment-emergent AEs are those with an o<br>and will be graded according to NCI CTCAE | onset on or after the initiation | of therapy, |
| Laboratory Data | Data will be summarized by: | | |
| | □ NCI-CTCAE for CTCAE-gradable parameters, and H/L for non-CTCAE-Gradable parameter | | |
| | ☐ H/L for all lab parameters | | |




### Tier 1 Study – Tables, Figures & Listings

| Standard TFLs | | | |
|---|---|---|---|
| Table No | Description | Variables/Analyses To Be Included | Subgroup Analyses |
| Table 1 | Summary of Patient Disposition | <ul> <li>Number of patients screened</li> <li>Number of patients randomized</li> <li>Number of patients treated</li> <li>Reason for treatment discontinuation</li> <li>Reason for study withdrawals</li> <li>Other, specify: Patient Deaths;</li> <li>Time on Study</li> </ul> | |
| Table 2 | Summary of Demographic<br>Characteristics | | |
| Table 3 | Summary of Disease History | <ul> <li>☐ Histology</li> <li>☐ Disease Staging</li> <li>☐ Time from Diagnosis</li> <li>☐ Other, specify: Baseline FISH</li> <li>Baseline</li> <li>Cytogenetics</li> </ul> | |
| Table 4 | Summary of Patient Treatment and Dose Modifications (reductions, interruptions) | | |
| Table 5 | Summary of Grade 3+ Adverse Events | | |
| Table 6 | Summary of Treatment-Related<br>Grade 3+ Adverse Events | | |
| Table 7 | Summary of Serious Adverse Events | | |
| Table 8 | Summary of Treatment-Related Serious Adverse Events | | |
| Table 9 | Summary of Treatment Related Adverse Events Leading to Death | | |
| Table 10 | Summary of Best Overall Response | | |
| Table 11 | Summary of Response Over Time | | |
| Table 12 | Summary of Progression-Free Survival (Kaplan-Meier estimates & 95 CI) | | |
| Table 13 | Summary of Overall Survival<br>(Kaplan-Meier estimates & 95 CI) | _ | |
| Table 14 | Summary of Adverse Events with >= 5% Frequency (for: CTGOV) | _ | |







REFERENCE SOP: CDS-0102

| Figure<br>No | Description | Variables/Analyses To Be Included | Subgroup Analyses |
|---|---|---|---|
| Figure 1 | Progression-Free Survival | Timescale to be used on horizontal axis: ☐ Day ☐ Week ☐ Month ☐ Year | |
| Figure 2 | Overall Survival | Timescale to be used on horizontal axis: ☐ Day ☐ Week ☐ Month ☐ Year | |
| • | | | |

| Listing<br>No. | Title | Variables/Analyses To Be<br>Included | Subgroup Analyses |
|---|---|---|---|
